CLINICAL TRIAL: NCT04124692
Title: A Randomized, Evaluator-blinded, No-treatment Controlled, Multicenter Study to Evaluate the Effectiveness and Safety of Sculptra Aesthetic for Correction of Cheek Wrinkles.
Brief Title: Safety and Effectiveness of Sculptra Aesthetic for Correction of Cheek Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USSA1812
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cheek Wrinkles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group: No-treatment (No Intervention): Participants will receive no treatment during the study.
- Treatment Group: Sculptra Aesthetic (Experimental): Participants will be injected with Sculptra Aesthetic by Treating Investigator at Day 1 until optimal correction achieved (up to 4 total treatment sessions)
  Interventions: Device: Sculptra Aesthetic new dilution

INTERVENTIONS:
Device: Sculptra Aesthetic new dilution — Treatment of cheek wrinkles
  Arms: Treatment Group: Sculptra Aesthetic

SUMMARY:
The study has been designed to evaluate the safety and effectiveness of Sculptra Aesthetic as a single regimen for correction of cheek wrinkles after changes in reconstitution and injection procedures compared to the approved label.

ELIGIBILITY:
Inclusion Criteria:

* Intent to undergo correction of cheek wrinkles on both sides of the face and a Galderma Cheek Wrinkles Scale (GCWS) At Rest score of Moderate or Severe on EACH side of the face.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any of the Sculptra Aesthetic constituents.
* Previous tissue augmenting therapy, contouring or revitalization treatment in the face, except the lips, with any of the following fillers prior to Baseline visit:

  1. Collagen, Hyaluronic Acid - 12 months
  2. Calcium Hydroxyapatite (CaHa), Poly L- Lactic Acid (PLLA) or permanent (nonbiodegradable)- Prohibited

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Galderma Research Site, Scottsdale, Arizona
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Redondo Beach, California
  - Galderma Research Site, San Diego, California
  - Galderma Research Site, Washington D.C., District of Columbia
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Alpharetta, Georgia
  - Galderma Research Site, New Orleans, Louisiana
  - Galderma Research Site, Rockville, Maryland
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Dallas, Texas
  - Galderma Research Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fabi SG, Le JHTD, Prygova I, Brasater D. Midface Projection Using Biostimulatory Poly- l -Lactic Acid Injectable Implant: A Subgroup Analysis of the Cheek Wrinkle Trial. Dermatol Surg. 2024 Dec 1;50(12):1137-1142. doi: 10.1097/DSS.0000000000004434. Epub 2024 Oct 17. PMID 39453400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 sites at the United States from 12 November 2019 to12 August 2021.
Pre-assignment Details: A total of 149 participants were enrolled and randomized, of which 97 received treatment and 52 received no treatment in this study.
Groups:
- Control Group: No-treatment: Participants received no treatment during the study.
- Treatment Group: Sculptra Aesthetic: Participants were injected with Sculptra Aesthetic by treating investigator at Day 1 until optimal correction achieved (up to 4 total treatment sessions).
Period: Overall Study
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Started | 52 | 97
Completed | 46 | 88
Not Completed | 6 | 9
Not completed — Medical reason | 0 | 1
Not completed — Withdrawal of informed consent (not due to coronavirus disease-19 concerns) | 2 | 1
Not completed — Withdrawal of informed consent (due to coronavirus disease-19 concerns) | 1 | 3
Not completed — Lost to Follow-up | 2 | 4
Not completed — Screen failure due to previous use of Radiesse | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who were randomized based on the treatment they were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic | Total
Number analyzed (Participants) | 52 | 97 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.72) | 60.9 (8.50) | 60.7 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 94 | 144
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 90 | 137
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 47 | 88 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fitzpatrick Skin Type score (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 2 | 4 | 6
    FST II | 18 | 25 | 43
    FST III | 21 | 47 | 68
    FST IV | 6 | 12 | 18
    FST V | 4 | 5 | 9
    FST VI | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the Galderma Cheek Wrinkles Scale (GCWS) at Rest at Month 12
Description: Responder rate was defined as the percentage of participants with at least a 1-grade improvement from baseline on the GCWS, on both sides of the face, concurrently. GCWS is a validated 5-point scale used to assess the severity of cheek wrinkles: 0 (none [no lines or wrinkles]), 1 (mild [only few superficial lines]), 2 (moderate [many superficial lines or a few shallow wrinkles]), 3 (severe [many shallow wrinkles or a few moderate depth wrinkles]) and 4 (very severe [many moderate wrinkles or at least one depth wrinkle with or without redundant folds]). Higher score means more severe (worse) wrinkles. The participant was to have a relaxed face during the assessment.
Time Frame: At Month 12
Population: ITT population included all participants who were randomized based on the treatment they were randomized to. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 46 | 88
percentage of participants | 26.1 | 71.6
Statistical Analysis 1: Comparison: Control Group: No-treatment vs Treatment Group: Sculptra Aesthetic; Test type: Superiority; p < 0.0001, Fisher Exact

2. Secondary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the GCWS at Rest at Months 7 and 9
Description: as for outcome 1
Time Frame: At Months 7 and 9
Population: ITT population included all participants who were randomized based on the treatment they were randomized to. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at the specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 45 | 85
percentage of participants
  Month 7: number analyzed (Participants) | 44 | 77
  Month 7 | 38.6 | 66.2
  Month 9 | 31.1 | 70.6
Statistical Analysis 1: Comparison: Control Group: No-treatment vs Treatment Group: Sculptra Aesthetic; Test type: Superiority; p = 0.0043, Fisher Exact
Statistical Analysis 2: Comparison: Control Group: No-treatment vs Treatment Group: Sculptra Aesthetic; Test type: Superiority; p < 0.0001, Fisher Exact

3. Secondary Outcome: Responder Rate Based on the Blinded Evaluator's Live Assessment of the GCWS Dynamic at Months 7, 9 and 12
Description: Responder rate was defined as the percentage of participants with at least a 1-grade improvement from baseline on the GCWS, on both sides of the face, concurrently. GCWS is a validated 5-point scale used to assess the severity of cheek wrinkles: 0 (none [no lines or wrinkles]), 1 (mild [only few superficial lines]), 2 (moderate [many superficial lines or a few shallow wrinkles]), 3 (severe [many shallow wrinkles or a few moderate depth wrinkles]) and 4 (very severe [many moderate wrinkles or at least one depth wrinkle with or without redundant folds]). Higher score means more severe (worse) wrinkles. The participant was to have a closed maximum smile during the assessment.
Time Frame: At Months 7, 9, and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 46 | 88
percentage of participants
  Month 7: number analyzed (Participants) | 44 | 77
  Month 7 | 27.3 | 67.5
  Month 9: number analyzed (Participants) | 45 | 85
  Month 9 | 22.2 | 64.7
  Month 12 | 28.3 | 70.5

4. Secondary Outcome: Percentage of Participants With Improvement Rate Based on the Independent Photographic Reviewer's Assessment
Description: Improvement rate based on the Independent Photographic Reviewer's assessment using random pairings of baseline and Month 12 photographs was done.
  An improved subject is defined as a subject for whom the Independent Photographic Reviewer identified the month 12 photograph in the pair as post-treatment.
Time Frame: At Month 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Control Group: No-treatment: Participants in this group received no treatment during the study.
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 44 | 84
percentage of participants
  Left Cheek | 29.5 | 53.6
  Right Cheek | 34.1 | 57.1

5. Secondary Outcome: Percentage of Participants With At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) Based on the Participants Live Assessment
Description: GAIS responder rates are based on independent assessments by the participant. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the participant to live assess the aesthetic improvement of the cheek wrinkles by responding to the question: "How would you describe the aesthetic improvement today compared to the photograph taken before treatment?" by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse.
Time Frame: At Months 7, 9, and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 46 | 88
percentage of participants
  Month 7: number analyzed (Participants) | 43 | 77
  Month 7 | 7.0 [1.5 to 19.1] | 93.5 [85.5 to 97.9]
  Month 9: number analyzed (Participants) | 44 | 85
  Month 9 | 6.8 [1.4 to 18.7] | 89.4 [80.9 to 95.0]
  Month 12 | 6.5 [1.4 to 17.9] | 92.0 [84.3 to 96.7]

6. Secondary Outcome: Percentage of Participants With At Least "Improved" on the GAIS Based on the Investigator Live Assessment
Description: GAIS responder rates are based on independent assessments by the investigator. Responder rate was defined as the percentage of participants with at least "Improved" when compared to baseline before first treatment. The 7-graded GAIS was used by the investigator to live assess the aesthetic improvement of the cheek wrinkles by responding to the question: "How would you describe the aesthetic improvement today compared to the photograph taken before treatment?" by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse.
Time Frame: At Months 7, 9, and 12
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 46 | 88
percentage of participants
  Month 7: number analyzed (Participants) | 44 | 77
  Month 7 | 6.8 [1.4 to 18.7] | 96.1 [89.0 to 99.2]
  Month 9: number analyzed (Participants) | 45 | 85
  Month 9 | 4.4 [0.5 to 15.2] | 92.9 [85.3 to 97.4]
  Month 12 | 4.3 [0.5 to 14.8] | 94.3 [87.2 to 98.1]

7. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look Younger?
Description: A 5-point subject satisfaction questionnaire with the following responses: Excellent, Very good, Good, Satisfactory, Not satisfied.
Time Frame: At Months 7, 9, and 12
Population: ITT population included all participants who were randomized based on the treatment they were randomized to. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints. The data was planned to be collected and analyzed for treatment group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 13
  At Month 7: Very good | 24
  At Month 7: Good | 15
  At Month 7: Satisfactory | 19
  At Month 7: Not satisfied | 6
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 19
  At Month 9: Very good | 26
  At Month 9: Good | 18
  At Month 9: Satisfactory | 15
  At Month 9: Not satisfied | 7
  At Month 12: Excellent | 15
  At Month 12: Very good | 29
  At Month 12: Good | 24
  At Month 12: Satisfactory | 11
  At Month 12: Not satisfied | 9

8. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Feel Better About Yourself?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 18
  At Month 7: Very Good | 20
  At Month 7: Good | 17
  At Month 7: Satisfactory | 18
  At Month 7: Not Satisfied | 4
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 18
  At Month 9: Very Good | 28
  At Month 9: Good | 22
  At Month 9: Satisfactory | 10
  At Month 9: Not Satisfied | 7
  At Month 12: Excellent | 21
  At Month 12: Very Good | 23
  At Month 12: Good | 27
  At Month 12: Satisfactory | 11
  At Month 12: Not Satisfied | 6

9. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Self-confidence?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 14
  At Month 7: Very good | 24
  At Month 7: Good | 16
  At Month 7: Satisfactory | 18
  At Month 7: Not Satisfied | 5
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 18
  At Month 9: Very good | 25
  At Month 9: Good | 25
  At Month 9: Satisfactory | 9
  At Month 9: Not Satisfied | 8
  At Month 12: Excellent | 20
  At Month 12: Very good | 21
  At Month 12: Good | 30
  At Month 12: Satisfactory | 10
  At Month 12: Not Satisfied | 7

10. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Overall Satisfaction With Your Appearance?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 17
  At Month 7: Very Good | 23
  At Month 7: Good | 13
  At Month 7: Satisfactory | 19
  At Month 7: Not Satisfied | 5
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 19
  At Month 9: Very Good | 28
  At Month 9: Good | 18
  At Month 9: Satisfactory | 13
  At Month 9: Not Satisfied | 7
  At Month 12: Excellent | 20
  At Month 12: Very Good | 21
  At Month 12: Good | 27
  At Month 12: Satisfactory | 13
  At Month 12: Not Satisfied | 7

11. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look/Feel More Confident in Your Life?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 19
  At Month 7: Very good | 19
  At Month 7: Good | 16
  At Month 7: Satisfactory | 18
  At Month 7: Not Satisfied | 5
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 17
  At Month 9: Very good | 26
  At Month 9: Good | 21
  At Month 9: Satisfactory | 15
  At Month 9: Not Satisfied | 6
  At Month 12: Excellent | 19
  At Month 12: Very good | 21
  At Month 12: Good | 28
  At Month 12: Satisfactory | 13
  At Month 12: Not Satisfied | 7

12. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look the Way You Feel?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 18
  At Month 7: Very good | 19
  At Month 7: Good | 12
  At Month 7: Satisfactory | 18
  At Month 7: Not Satisfied | 10
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 21
  At Month 9: Very good | 22
  At Month 9: Good | 22
  At Month 9: Satisfactory | 14
  At Month 9: Not Satisfied | 6
  At Month 12: Excellent | 19
  At Month 12: Very good | 20
  At Month 12: Good | 25
  At Month 12: Satisfactory | 17
  At Month 12: Not Satisfied | 7

13. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Firmness?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 18
  At Month 7: Very good | 24
  At Month 7: Good | 17
  At Month 7: Satisfactory | 13
  At Month 7: Not Satisfied | 5
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 25
  At Month 9: Very good | 26
  At Month 9: Good | 16
  At Month 9: Satisfactory | 11
  At Month 9: Not Satisfied | 7
  At Month 12: Excellent | 21
  At Month 12: Very good | 25
  At Month 12: Good | 26
  At Month 12: Satisfactory | 11
  At Month 12: Not Satisfied | 5

14. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Radiance?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 87
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 21
  At Month 7: Very good | 19
  At Month 7: Good | 13
  At Month 7: Satisfactory | 19
  At Month 7: Not Satisfied | 5
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 23
  At Month 9: Very good | 26
  At Month 9: Good | 13
  At Month 9: Satisfactory | 17
  At Month 9: Not Satisfied | 6
  At Month 12: Excellent | 22
  At Month 12: Very good | 23
  At Month 12: Good | 24
  At Month 12: Satisfactory | 10
  At Month 12: Not Satisfied | 8

15. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Improve Your Skin Sagging?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 15
  At Month 7: Very good | 23
  At Month 7: Good | 20
  At Month 7: Satisfactory | 7
  At Month 7: Not Satisfied | 12
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 23
  At Month 9: Very good | 19
  At Month 9: Good | 24
  At Month 9: Satisfactory | 11
  At Month 9: Not Satisfied | 8
  At Month 12: Excellent | 20
  At Month 12: Very good | 16
  At Month 12: Good | 32
  At Month 12: Satisfactory | 9
  At Month 12: Not Satisfied | 11

16. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make Your Skin Look More Refreshed?
Description: as for outcome 7
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Excellent | 16
  At Month 7: Very good | 23
  At Month 7: Good | 19
  At Month 7: Satisfactory | 12
  At Month 7: Not satisfied | 7
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Excellent | 23
  At Month 9: Very good | 26
  At Month 9: Good | 16
  At Month 9: Satisfactory | 14
  At Month 9: Not satisfied | 6
  At Month 12: Excellent | 23
  At Month 12: Very good | 21
  At Month 12: Good | 23
  At Month 12: Satisfactory | 14
  At Month 12: Not satisfied | 7

17. Secondary Outcome: Subject Satisfaction: Would You Say That the Treatment Results Are Natural Looking?
Description: A 5-point subject satisfaction questionnaire with the following responses: Strongly agree, Agree, Neither agree or Disagree, Disagree, Strongly disagree.
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Strongly agree | 47
  At Month 7: Agree | 25
  At Month 7: Neither Agree or Disagree | 4
  At Month 7: Disagree | 1
  At Month 7: Strongly Disagree | 0
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Strongly agree | 48
  At Month 9: Agree | 25
  At Month 9: Neither Agree or Disagree | 11
  At Month 9: Disagree | 0
  At Month 9: Strongly Disagree | 1
  At Month 12: Strongly agree | 47
  At Month 12: Agree | 30
  At Month 12: Neither Agree or Disagree | 7
  At Month 12: Disagree | 2
  At Month 12: Strongly Disagree | 2

18. Secondary Outcome: Subject Satisfaction: Would You Say the Subtle Changes Over Time Was Worth It?
Description: as for outcome 17
Time Frame: At Months 7, 9, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  At Month 7: number analyzed (Participants) | 77
  At Month 7: Strongly agree | 36
  At Month 7: Agree | 27
  At Month 7: Neither agree or Disagree | 11
  At Month 7: Disagree | 2
  At Month 7: Strongly disagree | 1
  At Month 9: number analyzed (Participants) | 85
  At Month 9: Strongly agree | 41
  At Month 9: Agree | 27
  At Month 9: Neither agree or Disagree | 13
  At Month 9: Disagree | 1
  At Month 9: Strongly disagree | 3
  At Month 12: Strongly agree | 41
  At Month 12: Agree | 31
  At Month 12: Neither agree or Disagree | 12
  At Month 12: Disagree | 2
  At Month 12: Strongly disagree | 2

19. Secondary Outcome: Subject Satisfaction: Would You Recommend the Treatment to a Friend?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: At Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  Yes | 78
  No | 10

20. Secondary Outcome: Subject Satisfaction: Would You do the Treatment Again?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: At Month 12
Population: ITT population included all participants who were randomized based on the treatment they were randomized to. Here, overall number of participants analyzed refer to the participants evaluated for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given timepoints. The data was planned to be collected and analyzed for treatment group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 88
Participants
  Yes | 76
  No | 12

21. Secondary Outcome: Change From Baseline in Satisfaction With Cheeks FACE-Q™ Questionnaire Rasch-transformed Total Scores
Description: The participant assessed satisfaction using the 5 questions on the FACE-Q: Satisfaction with Cheeks Appearance questionnaire measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, and 4=very satisfied. The responses to the items were converted to a 100-point Rasch transformed total score with 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A negative change from baseline indicates less improvement.
Time Frame: Treatment group: Baseline, Months 1, 2, 3, 7, 9 and 12; Control group: Baseline, Months 7, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 45 | 94
score on a scale
  At Month 1: number analyzed (Participants) | 0 | 94
  At Month 1 |  | 21.3 (24.25)
  At Month 2: number analyzed (Participants) | 0 | 87
  At Month 2 |  | 31.6 (28.45)
  At Month 3: number analyzed (Participants) | 0 | 81
  At Month 3 |  | 38.6 (26.51)
  At Month 7: number analyzed (Participants) | 42 | 77
  At Month 7 | -4.1 (20.34) | 38.6 (26.30)
  At Month 9: number analyzed (Participants) | 44 | 85
  At Month 9 | -3.6 (21.36) | 37.9 (26.63)
  At Month 12: number analyzed (Participants) | 45 | 88
  At Month 12 | -3.6 (21.76) | 40.0 (29.07)

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs with a start date on or after the first dose of investigational product or a start date before the date of the first dose of investigational product that increased in severity or after the date of the first dose. A SAE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, and was an important medical event. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to end of the study (up to Month 12)
Population: Safety population (SP) included all participants who were treated with Sculptra Aesthetic or randomized to the no treatment control group.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: No-treatment: Participants were injected with Sculptra Aesthetic by treating investigator at Day 1 until optimal correction achieved.
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
Number analyzed (Participants) | 52 | 97
Participants
  Non-serious AE | 3 | 43
  Serious AE | 0 | 3

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of the study (up to Month 12)
Description: SP included all participants who were treated with Sculptra Aesthetic or randomized to the no treatment control group.
Groups:
- Treatment Group: Sculptra Aesthetic: Participants were injected with Sculptra Aesthetic by treating investigator at Day 1 until optimal correction achieved.
Arm/Group | Control Group: No-treatment | Treatment Group: Sculptra Aesthetic
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/52 | 3/97
Other Adverse Events (participants affected / at risk) | 0/52 | 11/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group: No-treatment (N=52) | Treatment Group: Sculptra Aesthetic (N=97)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Obstruction gastric and small intestine adenocarcinoma (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group: No-treatment (N=52) | Treatment Group: Sculptra Aesthetic (N=97)
Injection site bruising (General disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT04124692/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT04124692/SAP_001.pdf